CLINICAL TRIAL: NCT07354828
Title: Optimization and Validation of Quality Control Indicators for Coronary Revascularization Based on Antiplatelet Therapy: Establishment of a Quality Control Standard System for Coronary Revascularization in Coronary Heart Disease Based on Dual Antiplatelet Therapy (DAPT)
Brief Title: Optimization and Validation of Quality Control Indicators for Coronary Revascularization Based on Antiplatelet Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director, clinical professor, Shenyang Northern Hospital
Other Study IDs: 2025ZD0546702
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome (ACS); High Bleeding Risk (HBR); Coronary Artery Disease (CAD)
Keywords: Dual Antiplatelet Therapy (DAPT); Acute Coronary Syndrome (ACS); High Bleeding Risk (HBR); Percutaneous Coronary Intervention (PCI); OPT-CAD Score; Quality Control Indicators; Coronary Revascularization; Prospective Cohort Study; Real-World Research; Bleeding Events; Ischemic Events; Medication Adherence; Post-PCI Prognosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Ischemic Risk (OPT-CAD < 90): This group includes patients with high bleeding risk (meeting ARC-HBR criteria) who are diagnosed with Acute Coronary Syndrome (ACS) and have undergone Percutaneous Coronary Intervention (PCI) with at least one Drug-Eluting Stent (DES) implantation. All participants have an OPT-CAD score < 90, indicating low ischemic risk. They receive routine Dual Antiplatelet Therapy (DAPT) for 6-12 months as per clinical guidelines (specific regimens determined by attending physicians). During the 12-month follow-up, data on DAPT adherence, discontinuation reasons, and clinical outcomes (bleeding/ischemic events, mortality) will be collected to compare with the moderate/high ischemic risk group.
- Moderate/High Ischemic Risk (OPT-CAD ≥ 90): This group comprises patients who meet the same baseline criteria as Group 1: high bleeding risk (ARC-HBR positive), ACS diagnosis, PCI with DES implantation, and ability to tolerate 12-month DAPT. The key distinction is an OPT-CAD score ≥ 90, classifying them as moderate/high ischemic risk. They also receive standard 6-12 month DAPT (regimens decided by clinicians). Follow-up procedures and data collection are identical to Group 1, aiming to verify the predictive value of the OPT-CAD score by comparing clinical outcomes between the two groups.

SUMMARY:
Study Purpose Coronary heart disease (CAD) is a leading global cause of death, with Acute Coronary Syndrome (ACS) as its acute and life-threatening subtype. Percutaneous Coronary Intervention (PCI) plus stent implantation is the first-line treatment for ACS, and post-PCI Dual Antiplatelet Therapy (DAPT, aspirin + P2Y₁₂ inhibitor) is core for thrombosis prevention but increases bleeding risk. Approximately 40% of ACS patients are classified as High Bleeding Risk (HBR). China lacks a unified DAPT quality control system, and the predictive value of the OPT-CAD ischemic risk score for this population remains unvalidated. This study aims to: 1) Evaluate the feasibility and influencing factors of the DAPT quality control system in HBR ACS patients post-PCI; 2) Verify the accuracy of the OPT-CAD score in predicting ischemic risk, providing evidence for personalized treatment.

Eligibility Criteria Inclusion Criteria Aged ≥18 years; Diagnosed with ACS and implanted with at least one drug-eluting stent (DES) during PCI; Meets ARC-HBR (Academic Research Consortium for High Bleeding Risk) HBR definition (1 major criterion or 2 minor criteria); Able to complete OPT-CAD scoring; Tolerates 12-month DAPT (physician assessment); Signs informed consent. Exclusion Criteria Allergy to aspirin, clopidogrel, ticagrelor, or other study-related antiplatelet drugs; Severe ischemia or major bleeding during current hospitalization; Terminal illness with life expectancy <1 year; Pregnant or planning pregnancy within 1 year; Enrolled in other ongoing clinical studies. Study Process

This is a multi-center prospective cohort study (we will follow eligible patients over 12 months to collect real-world data without changing their standard care) recruiting 3,500 participants nationwide. Post-enrollment:

Receive 6-12 months of standard DAPT (regimen determined by your physician); Follow-ups at 1 month (±7 days), 3 months (±14 days), 6 months (±30 days), and 12 months (±30 days) post-PCI (via phone or outpatient visit) to collect medication adherence, bleeding/ischemic events, and clinical outcomes; Confidential data collection via a secure Electronic Data Capture (EDC) system. Study Endpoints Primary Endpoints Feasibility of the DAPT quality control system, inter-hospital differences in DAPT use, 6-12 month DAPT completion rate, and impact of DAPT interruption on patient outcomes; Accuracy of the OPT-CAD score in predicting ischemic risk for HBR patients. Secondary Endpoints 12-month bleeding event rates (BARC 1-5 types, including minor bleeding like puncture site bleeding and major bleeding like intracranial hemorrhage); 12-month ischemic event rates (including target lesion failure-cardiac death, target vessel-related myocardial infarction, or target lesion revascularization-all-cause death, ischemic stroke, definite stent thrombosis, etc.); DAPT interruption rate, P2Y₁₂ inhibitor discontinuation rate (≥1 week), and aspirin discontinuation rate (≥1 week).

Key Information for Participants Voluntary participation: You may withdraw anytime without penalty or loss of medical benefits; Confidential data protection: Personal information will be anonymized with a unique study ID; Free study-related assessments and follow-ups; Prompt medical care will be provided for any adverse events. For inquiries, contact the study team at the participating hospital.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, observational registry cohort study designed to evaluate real-world dual antiplatelet therapy (DAPT) management in high-bleeding-risk patients with acute coronary syndrome (ACS) undergoing percutaneous coronary intervention (PCI).

Eligible patients undergoing PCI will be screened against the study inclusion and exclusion criteria. Patients who meet eligibility requirements will be invited to participate, provide informed consent, and be assigned a unique study identification number. Study participation will not alter routine clinical care, and all treatment decisions, including DAPT regimen selection and duration, will be determined by the treating physician in accordance with standard clinical practice.

A total of approximately 3,500 evaluable patients are planned to be enrolled across multiple centers nationwide, including prefecture-level/district/county hospitals and provincial or national key hospitals. Enrollment will reflect real-world clinical practice, with no more than a predefined proportion of patients enrolled at any single site.

Clinical data will be collected prospectively at baseline and during routine follow-up at approximately 1, 3, 6, and 12 months following PCI. Collected information will include patient characteristics, PCI-related data, DAPT treatment patterns, and clinical outcomes.

The registry is designed to characterize real-world application of a DAPT quality control indicator system and to evaluate the prognostic performance of the OPT-CAD score in high-bleeding-risk ACS patients. Findings from this study are expected to provide real-world evidence to support standardized DAPT quality control and personalized antiplatelet therapy in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Clinically diagnosed with ACS and received implantation of at least one drug-eluting stent (DES)
* Meets 1 major criterion or 2 minor criteria of the ARC-HBR high-bleeding-risk definition
* Able to complete the OPT-CAD score calculation
* Judged by the investigator to tolerate DAPT for at least 12 months
* Signed the informed consent form

Exclusion Criteria:

* Allergy to study medications such as aspirin, clopidogrel, or ticagrelor
* Occurrence of major ischemic or bleeding events during the current hospitalization
* Presence of other severe diseases with a life expectancy of less than one year
* Pregnancy, or women of childbearing potential who plan to become pregnant within one year
* Current participation in another clinical study and still within its observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from inpatients admitted to multiple nationwide medical centers (including prefecture/county-level hospitals and provincial/national key hospitals) who are clinically diagnosed with Acute Coronary Syndrome (ACS) and undergo Percutaneous Coronary Intervention (PCI) with Drug-Eluting Stent (DES) implantation during hospitalization. The source population consists of ACS patients who meet the clinical diagnostic criteria, require PCI treatment, and are potentially at high bleeding risk (may fulfill ARC-HBR criteria). Patients with clear contraindications to Dual Antiplatelet Therapy (DAPT), inability to complete follow-up, or other conditions that make them unsuitable for the study are excluded from the source population.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The overall composite of 11 performance measures for DAPT-based Quality Control Standard System for Coronary Artery Disease Revascularization. | 12 months
  The proportion of ACS patients scheduled for stent implantation during PCI who undergo risk stratification; The proportion of ACS patients undergoing PCI who initiate DAPT during the procedure; The proportion of ACS patients who maintain DAPT for at least 12 months after PCI; In patients at "high bleeding risk", the proportion of patients whose DAPT regimens are adjusted according to risk; The proportion of patients with implanted BRS who maintain DAPT for more than 12 months; The proportion of patients receiving alternative DAPT regimens due to drug intolerance or allergy; The proportion of implementation of optimized regimens combining anticoagulation with DAPT; The proportion of DAPT adjustment following bleeding events; Incidence of ischemic events: cardiac death, ischemic stroke, definite stent thrombosis, TVR, and TLF; Incidence of bleeding events: BARC Types 3/5 bleeding; The proportion of patients adherent to standardized DAPT.
Accuracy of the OPT-CAD score in predicting ischemia risk in high-bleeding-risk patients. | 12 months
  The OPT-CAD score (Optimal antiPlatelet Therapy for Chinese patients with Coronary Artery Disease) is an ischemic risk scoring system developed based on the Chinese OPT-CAD registry study (107 centers, 14,032 patients). It is specifically used to predict long-term ischemic events and all-cause mortality in Chinese patients with coronary artery disease, especially those with acute coronary syndrome (ACS). OPT-CAD score ranges from 0 to 257 points in total. Patients are divided into three risk levels based on their total scores, corresponding to different incidences of ischemic events:Low risk 0-90 points ;Medium risk 91-150 points High risk ≥151 points.

SECONDARY OUTCOMES:
Incidence of first BARC 3/5 bleeding within 12 months; | 12 months
  Incidence rate of major bleeding events (Bleeding Academic Research Consortium (BARC)[1] defined Type 3 and Type 5 bleeding) [1]Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. PMID: 21670242.
Incidence of first BARC 2/3/5 bleeding within 12 months | 12 months
  Incidence rate of bleeding events (Bleeding Academic Research Consortium (BARC)[1] defined Type2, Type 3 and Type 5 bleeding, including puncture site bleeding, gastrointestinal bleeding, and intracranial hemorrhage.)[1]Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. PMID: 21670242.
Incidence of first BARC 1/2/3/5 bleeding within 12 months | 12 months
  Incidence rate of bleeding events (Bleeding Academic Research Consortium (BARC)[1] defined Type1, Type2, Type 3 and Type 5 bleeding, including puncture site bleeding, gastrointestinal bleeding, and intracranial hemorrhage.)[1]Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. PMID: 21670242.
Incidence of target lesion failure (TLF) within 12 months | 12 months
  defined as cardiac death, target vessel myocardial infarction, and target lesion revascularization
Incidence of different types of ischemic events within 12 months | 12 months
  * All-cause death
  * Cardiac death
  * Ischemic stroke
  * Definite stent thrombosis
  * Target vessel revascularization
Discontinuation rate of continuous dual antiplatelet therapy; | 12 months
Discontinuation rate of P2Y12 inhibitor | 12 months
  discontinuation for ≥1 week
Discontinuation rate of aspirin | 12 months
  discontinuation for ≥1 week

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Li PX.Long-term prognosis and influencing factors of high bleeding risk ACS patients after PCI [Master's Thesis]; 2023.2.Yin P,Qi JL,Liu YN,et al.China's disease burden study report 2005-2017.Chinese Circulation Journal 2019; 34(12):1145-1154.3.Liu MB,He XY,Yang XH,et al. Summary of "China Cardiovascular Health and Disease Report 2023"(Epidemiology of cardiovascular diseases and interventional diagnosis and treatment status). Chinese Journal of Interventional Cardiology 2024;32(10): 541-550.4.Tan MQ,Yin CE,Wang FJ.Interpretation of the 2018 updated universal definition of myocardial infarction.Journal of Practical Electrocardiology 2018; 27(06):381-385.